CLINICAL TRIAL: NCT06084741
Title: Omitting of Usage of Intraabdominal Drains After Repair of Peptic Ulcer Perforations Compared to Traditional Use of Drains; Comparative Study
Brief Title: Omitting Drains After Repair of Peptic Ulcer Perforations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elshwadfy Nageeb, Lecturer of general surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-79-2023
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Peptic Ulcer Perforations
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain group (Active Comparator): In Group A the investigators will put intraabdominal drains
  Interventions: Other: Using intraabdominal drains
- No drain group (Experimental): The investigators will not put any intraabdominal drains
  Interventions: Other: Omitting of usage of intraabdominal drains after repair of peptic ulcer perforations

INTERVENTIONS:
Other: Omitting of usage of intraabdominal drains after repair of peptic ulcer perforations — omitting the intraabdominal drains
  Arms: No drain group
Other: Using intraabdominal drains — The investigators will put intraabdominal drains
  Arms: Drain group

SUMMARY:
. This study aimed to evaluate ERAS application outcomes via omitting the intraabdominal drains compared to regular using of the drains in patients undergoing perforated duodenal ulcer repairs in emergency abdominal surgeries.

DETAILED DESCRIPTION:
Patients will be randomly assigned into two groups. In Group A : the investigators will put intraabdominal drains, and in Group ,thd investigators will not put any intraabdominal drains. Our primary outcomes will be hospital stayl engthand pain score;Data analysis packages will be SPSS version 21 Qualitative data will be presented by number and percentage, quantitative data by mean, standard deviation, median and interquartile range.

ELIGIBILITY:
Inclusion Criteria:

- Patients older than 18 years with perforated peptic ulcer who underwent exploratory laparotomy or laparoscopy and repair with omental pedicle techniques will included in the study.

Exclusion Criteria:

* preoperative shock on admission.

  * Delayed presentation more than 24 hours.
  * known malignant gastric ulcers confirmed by histopathology.
  * the presence of neuropsychiatric disease, pregnant and lactating women.
  * predisposing factors for impaired wound healing (e.g., currently using immunosuppressive agents, or chronic use of steroids), the presence of HIV/AIDS.
  * Intraoperative findings consistent with malignant ulcers. • American Society of Anesthesiologists grade III/IV, or had an alternative perioperative diagnosis. • Ulcer size more than 2 cm in diameter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
number of days of hospital stay | Up to 30 days
  hospital stay length
number of patients with infection-related postoperative complications such as superficial, deep or organ space SSI, hospital acquired pneumonia | 30 days
  number of patients with infection-related postoperative complications such as superficial, deep or organ space SSI, hospital acquired pneumonia
incidence of Post operative repair leak | 30 days
  incidence of Post operative repair leak

SECONDARY OUTCOMES:
number of days before frist bowel motion | 7 days
  number of days before frist bowel motion
severity of operative pain measured by Visual Analogue Scale (VAS | 7 days
  from 1 to 10 1 indicated minimum pain and 10 maximum pain
INCIDENCE OF postoperative nausea and vomiting (PONAV | 7 days
  INCIDENCE OF postoperative nausea and vomiting (PONAV

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed ElShwadfy, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nageeb ME, Tobar W, Saqr A, Ragab AA, Elansary AMSEO. No drains versus drains after perforated peptic ulcer repair: A randomized controlled trail. Eur J Trauma Emerg Surg. 2024 Oct;50(5):2137-2145. doi: 10.1007/s00068-024-02551-6. Epub 2024 Jun 15. PMID 38878063